CLINICAL TRIAL: NCT06915922
Title: Therapeutic Neodymium-doped Yttrium-Aluminum-Garnet (Nd:YAG) Laser Vitreolysis for Vitreous Floaters - A Study to Quantify Visual Quality of Life, Vitreous Structure, and Vision Before and After Nd:YAG Laser Vitreolysis in Patients With Vision Degrading Myodesopsia
Brief Title: YAG Laser Vitreolysis for Vitreous Floaters
Acronym: YLV Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VMR Consulting, Inc. (Other)
Collaborators: Quantel Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023000367
Record Dates: First submitted 2025-03-26; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Posterior Vitreous Detachment; Myopic Vitreopathy; VISION DEGRADING MYODESOPSIA
MeSH Terms: conditions — Vitreous Detachment | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neodymium-doped Yttrium-Aluminum-Garnet (Nd:YAG) Laser Vitreolysis (Other)
  Interventions: Device: Neodymium-doped yttrium-aluminum-garnet (Nd:YAG) laser therapy

INTERVENTIONS:
Device: Neodymium-doped yttrium-aluminum-garnet (Nd:YAG) laser therapy — Nd:YAG laser treatment(s) for Vision Degrading Myodesopsia (clinically significant vitreous floaters) in eyes with vitreous opacities due to myopic vitreopathy and posterior vitreous detachment (PVD).

SUMMARY:
The purpose of this study is to measure how the quality of life, the structure of eye, and vision change after treatment for the opacities in the gel (vitreous) that fills the center of eye which cause vision disturbances commonly called "floaters".

In this study the vitreous floaters are treated using a Neodymium-doped yttrium-aluminum-garnet (Nd:YAG) laser. The FDA has approved the use of this laser to treat membranes in the eye.

ELIGIBILITY:
Inclusion Criteria:

* Only one eye per patient will be included in this study
* Able and willing to give informed consent
* Age ≥18 years
* Suffering from symptomatic vitreous floaters
* Floaters arising from either/both:

  * myopic vitreopathy
  * posterior vitreous detachment
* Floaters meeting the following characteristics:

  * Present for ≥3 months
  * One single or more dense and well-defined vitreous opacities,
  * A Weiss Ring or opacities which are within the safety area, at least 3mm away from the retina and 6mm away from the lens
  * Visible on contact lens biomicroscopy

Exclusion Criteria:

* Patient presenting with vitreous opacities outside of the described safety area (within 3mm of the retina or 6mm from the lens)
* Have clinically significant cataract (lens opacification) in one or both eyes which are in the opinion of the examining doctor more significant in impacting vision as compared to that caused by vitreous opacities; or cataract expected to need cataract surgery during the duration of the study
* Present with untreated retinal tears or retinal holes requiring treatment at the discretion of the study investigator
* Have high risk of peripheral lesions requiring treatment at the discretion of the study investigator
* Have synchysis scintillans (unusual vitreous opacities from old blood)
* Have asteroid hyalosis (unusual vitreous opacities from cholesterol)
* Have vitreous hemorrhage (fresh blood in the center of the eye)
* Have active photopsia (flashing lights)
* History of previous YAG laser vitreolysis treatments, or vitrectomy for any condition (retinal detachment, proliferative diabetic retinopathy, etc.)
* Have Posterior Vitreous Detachment (separation of vitreous away from the retina lining the inside of the back of the eye) within the past 3 months
* Are unable to attend study appointments
* Have any other significant ocular or non-ocular condition that, at the discretion of the study investigator, puts the subject at risk or influences the results of the study
* History of intraocular surgery within 6 months from study entry
* History of retinal laser within 2 months from study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Measures of vitreous structure by quantitative ultrasonography | baseline, 3 months, 6 months, 12 months

SECONDARY OUTCOMES:
Measures of visual function using contrast sensitivity | baseline, 3 months, 6 months, 12 months
Evaluation of quality of life using Visual Function Questionnaire (VFQ-25) | baseline, 3 months, 6 months, 12 months
  Individual scores (NEI VFQ 25 score) are recoded and transformed on a scale from 0 to 100, where 100 represents the best possible performance and 0 represents the worst
Evaluation of quality of life using Vitreous Floater Functional Questionnaire (VFFQ) | baseline, 3 months, 6 months, 12 months
  Individual scores (VFFQ score) are recoded and transformed on a scale from 0 to 100, where 100 represents the best possible performance and 0 represents the worst
Evaluation of Visual Acuity (ETDRS LogMAR) | baseline, 3 months, 6 months, 12 months
Evaluation of Near Visual Acuity | baseline, 3 months, 6 months, 12 months
Evaluation of retinal electrical activity changes in response to light stimuli (Photopic Negative Response amplitude) using Electroretinography (ERG) | baseline, 3 months, 6 months, 12 months
Visual evaluation of retinal structure changes in sagittal mode using optical coherence tomography (OCT) centered on the fovea | baseline, 3 months, 6 months, 12 months
Evaluation of central visual field changes (median light sensitivity) using microperimetry | baseline, 3 months, 6 months, 12 months
  Scale 0-36dB (0 worst condition; 36dB the best condition)

CONTACTS AND LOCATIONS:
Locations (1):
- VMR Institute for Vitreous Macula Retina, Huntington Beach, California, United States